CLINICAL TRIAL: NCT03357432
Title: Determining Whether Gelatin, Hydrolyzed Collagen and Gelatin/Collagen Mixture Have Similar Effects on Collagen Synthesis
Brief Title: Gelatin, Collagen, Gummy and PINP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 1140867
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Collagen Synthesis
Keywords: collagen; gelatin; PINP
MeSH Terms: interventions — Gelatin; Collagen

STUDY DESIGN:
Intervention Model Description: A crossover design where subject are randomized to consume all 3 intervention doses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- effects of gelatin, collagen on PINP levels (Experimental): The study is aimed at determining if the same dose of gelatin, hydrolyzed collagen (administered in a beverage form) or a mixture gelatin/hydrolyzed collagen (administered in a gummy form) with a standard dose of vitamin C (50 mg) has a similar effect a marker of collagen synthesis (PINP). In a randomized, crossover design subjects consume 3 different nutritional supplements: (a) 15 of gelatin, (b) 15 hydrolyzed collagen (administered in a beverage form) or (c) 15 g of gelatin/hydrolyzed collagen mixture all with a standard dose of vitamin C (50 mg) 1 hour prior to exercise stimulus (6 minutes of jump rope). A baseline assessment with only the jump rope and no intervention will also be conducted prior to the interventions. Each intervention will be separated by a >24 hr washout. Following completion of exercise, subjects will remain in the lab in a rested state for the subs
  Interventions: Other: gelatin, collagen, gummy dose

INTERVENTIONS:
Other: gelatin, collagen, gummy dose — The study is aimed at determining if the same dose of gelatin, hydrolyzed collagen (administered in a beverage form) or a mixture gelatin/hydrolyzed collagen (administered in a gummy form) with a standard dose of vitamin C (50 mg) has a similar effect a marker of collagen synthesis (PINP). In a randomized, crossover design subjects consume 3 different nutritional supplements: (a) 15 of gelatin, (b) 15 hydrolyzed collagen (administered in a beverage form) or (c) 15 g of gelatin/hydrolyzed collagen mixture all with a standard dose of vitamin C (50 mg) 1 hour prior to exercise stimulus (6 minutes of jump rope). A baseline assessment with only the jump rope and no intervention will also be conducted prior to the interventions. Each intervention will be separated by a >24 hr washout. Following completion of exercise, subjects will remain in the lab in a rested state for the subsequent 4 hours. After 4 hours blood samples will be collected. Blood samples will be used for PINP analysis.

SUMMARY:
Previous work has shown that gelatin supplementation could increase collagen synthesis in humans. In this study subjects consume placebo, 5 or 15 g of gelatin with a standard amount of vitamin C (48 mg) 1 hour before 6 minutes of jump rope exercise. The feeding and exercise intervention was repeated every 6 hours while the subjects were awake for three days and the amount of the amino terminal procollagen I peptide (PINP) was determined; a marker of collagen synthesis, in the blood. Consistent with the hypothesis that gelatin increases collagen synthesis in humans; the amount of PINP in the 15 g gelatin group was significantly higher than either the placebo or the 5 g groups. These data conclusively demonstrate that gelatin supplementation can increase exercise-induced collagen synthesis in humans. Hydrolyzed collagen has a similar amino acid profile, in particular with high concentrations of glycine, proline, hydroxyproline, and arginine. Thus, the current study aims to determine is the same dose of gelatin, hydrolyzed collagen and a gelatin/collagen mix, all with a standard dose of vitamin C effect PINP levels similarly.

DETAILED DESCRIPTION:
In preliminary work investigating the physiological determinants of maximal performance in throwing events, researchers found that the best predictor of elite performance was the rate of force development (RFD; Force (N) x time (sec)) when performing and isometric squat. Therefore, it is not surprising that in order to maximize performance, athletes train to optimize RFD.

RFD is determined by three factors:

1. Neural activation of the muscles
2. Type of motor protein (fast or slow myosin)
3. Force transfer Interestingly, performance in power movements (that are highly dependent on RFD) like vertical jump is closely related to tendon stiffness and inversely related to muscle size. This indicates that force transfer, in the form of tendon stiffness, plays an important role in performance and can explain a large amount of variance in determining an athlete's ability to rapidly develop force during a dynamic movement.

The stiffness of a tendon is determined by the amount and cross-linking of collagen within the tissue. Acute exercise is known to increase collagen synthesis as well as the expression of the primary enzyme involved in collagen cross-linking, lysyl oxidase. The result is a denser and stiffer tissue after training. Even though the relationship between exercise and collagen synthesis is known, whether this measure of performance can be improved with nutritional interventions has not been determined.

A recent study looking at amino acid levels following consumption of increasing doses of gelatin (derivative of collagen) in human subjects has shown that the key primary and trace amino acids found in collagen increase in human serum after consuming gelatin. Further, the peak of these amino acids occurs 60 minutes after consuming the gelatin supplement. Therefore, consuming a collagen supplement 1 hour before an exercise intervention should maximize delivery of amino acids to bone and other connective tissues.

To determine whether the gelatin supplement could increase collagen synthesis in humans, subjects consumed placebo, 5 or 15 g of gelatin with a standard amount of vitamin C (48 mg) 1 hour before 6 minutes of jump rope exercise. The feeding and exercise intervention was repeated every 6 hours while the subjects were awake for three days and the amount of the amino terminal procollagen I peptide (PINP) was determined; a marker of collagen synthesis, in the blood. Consistent with the hypothesis that gelatin increases collagen synthesis in humans; the amount of PINP in the 15 g gelatin group was significantly higher than either the placebo or the 5 g groups. These data conclusively demonstrate that gelatin supplementation can increase exercise- induced collagen synthesis in humans.

Similarly, supplementation with collagen hydrolysate has previously been shown to improve cartilage function in a randomized clinical trial in patients with osteoarthritis [9]. McAlindon and colleagues showed that consuming 10 g of collagen hydrolysate per day resulted in an increase in gadolinium enhanced MRI of collagen [9]. This finding suggests that the hydrolyzed collagen increased cartilage formation. In agreement with this finding, a 24- week randomized clinical trial in athletes showed that 10 g of GELITA® collagen hydrolysate significantly decreased knee pain. Mouse studies using C14 labeled hydrolyzed collagen hydrolysate demonstrated that >95% of the hydrolyzed collagen was absorbed in the first 12 hours after feeding. Interestingly, even though tracer from a separate C14 labeled proline could be incorporated into skin collagen at the same rate as tracer from hydrolyzed collagen, tracer from the hydrolyzed collagen was incorporated into the collagen of cartilage and muscle two-fold more than the tracer from proline. These data suggest that musculoskeletal collagen synthesis is greater in response to gelatin or hydrolyzed collagen than to the individual amino acids.

Even though the blood measure of PINP levels likely reflects bone collagen synthesis, using an engineered ligament model, a similar response has been demonstrated in tendons/ligaments treated with serum from people 1 hour after supplementation with gelatin. This work has shown that in the presence of serum isolated from the 5 and 15 grams of gelatin groups a step-wise increase in the collagen content of the ligaments. From this work, it can be ascertained that PINP can be used dependably as an indirect marker of collagen synthesis and that the changes observed in bone (blood levels) reflect what is occurring in other connective tissues as well.

The current study aims to determine if the same dose (15 g) of gelatin, hydrolyzed collagen and a mixture of gelatin and hydrolyzed collagen in a gummy form, all with a standard dose of vitamin C (50 mg) have a similar effect on PINP levels; an indirect marker of collagen synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active male athletes between the ages of 18-50 years of age training 5-6 days per week including at least 1 training session of running per week.

Exclusion Criteria:

* Receiving any medication that may interfere with the study.
* History of more than 3 musculoskeletal injuries within the past 12 months.
* Health or dietary restriction that would be affected by the supplementation protocol.
* The initial phases of this study will be performed in males since collagen synthesis varies significantly throughout the menstrual cycle in females. Since collagen is the main outcome measure for this study this natural variation would confound the initial phase of the work. Provided this work proves successful then we will aim to process with similar research in females.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male healthy active
Enrollment: 11 (Actual)
Dates: Start 2017-10-21 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
PINP levels | 4 weeks
  To determine optimal dose of supplemental hydrolyzed collagen and vitamin C required to maximally elevate PINP levels (a marker of collagen synthesis) in healthy athletes.

CONTACTS AND LOCATIONS:
Locations (1):
- Biological Sciences, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No